CLINICAL TRIAL: NCT05473923
Title: Study on Precision Treatment Strategy Through PTCs (patient-derived Tumor-like Cell Clusters)-based Drug Screening for Recurrent High-grade Gliomas
Brief Title: PTCs-based Precision Treatment Strategy on Recurrent High-grade Gliomas
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing GeneX Health Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Yang Zhang, Ph.D. & M.D., Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-069-02
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Recurrent High Grade Glioma
Keywords: precision medicine; organoid-based drug screening; bioinformatic prediction for drug response
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Receiving chemotherapeutic or targeted drugs recommended by molecular tumor board. (Experimental): These drugs included all the FDA-approved drugs that have been used in treating gliomas. A single drug or a drug combination for a specific patient will be recommended by the molecular tumor board, comprising neurooncologists, neurosurgeons, pharmacologists, cancer biologists, radiologists and bioinformaticians, will recommend , based on their expertise, patients willingness as well as evidences from PTCs-drug screening and bioinformatic prediction for drug response.
  Interventions: Drug: Receiving chemotherapeutic or targeted drugs recommended by molecular tumor board.

INTERVENTIONS:
Drug: Receiving chemotherapeutic or targeted drugs recommended by molecular tumor board. — Patients will be treated with FDA-approved chemotherapeutic or targeted drugs which were recommended by the molecular tumor board (MTB), based on their expertise, patients willingness as well as evidences from PTCs-drug screening and bioinformatic prediction for drug response.

SUMMARY:
This trial is an open-label, single-arm, phase 0/1 study of high-grade glioma that aims to evaluate the feasibility, preliminary efficacy and safety of the precision treatment strategy.

DETAILED DESCRIPTION:
The investigators have established a precision treatment strategy, that select chemotherapeutic drugs or targeted drugs based on information from PTCs drug-screening or/and bioinformatic prediction. In this study, the investigators are going to exploit this strategy for the precision treatment of recurrent high-grade gliomas. The investigators will evaluate the feasibility, safety and preliminary efficacy via collecting the indexes comprising clinical presentation, results of imaging examination, clinical assays, KPS, neurological score, etc.

ELIGIBILITY:
Inclusion Criteria:

* 1 At the age of 18~75, regardless the gender
* 2 The lesion of primary surgery was diagnosed as WHO II~IV Glioma by histologic pathology
* 3 Received radiotherapy and Temozolomide-based chemotherapy within 5 years
* 4 Recurrent and respectable gliomas, and have been neurosurgically resected
* 5 The resected recurrent gliomas was identified as WHO III~IV Glioma by histologic pathology
* 6 None postoperative standard therapeutic regimens can be followed when participating the recruitment
* 7 Can understand the trial's content and sign informed consent

Exclusion Criteria:

* 1 Having other untreated malignant tumors
* 2 The amount of resected tumors is not enough for genomic sequencing or PTCs drug screening
* 3 Received Carmustine implants within 6 months prior to enrollment
* 4 Subjects with active HBC, HCV or HIV infection
* 5 Subjects with uncontrolled cardio- or cerebro- vascular diseases
* 6 Subjects with uncontrolled psychiatric diseases or condition that could increase adverse events or interfere the evaluation of outcomes
* 7 Subjects with other conditions in their active phase that would interfere trial participation
* 8 Subjects receiving immunosuppressants after organ transplantation
* 9 Subjects with unstable pulmonary embolism, deep venous embolism, or other major arterial and venous thromboembolic events that occur within 30 days before the enrollment, or receiving anticoagulant therapy
* 10 Subjects in pregnancy or breastfeeding, or those who plan to become pregnant during treatment or within 2 months after the end of treatment
* 11 Subjects with other conditions that would interfere participating in the trial at the investigator's discretion
* 12 Subjects with medical conditions that affect signing the written informed consent or complying with the research procedures; or patients who are unwilling or unable to comply with the research procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who accomplish the recommended regimen for at least 1 course. | 24 months

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs) | From the first shot to 4 weeks after the last shot
  AEs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Ratio of 6 months overall survival (OS) | 6 months
  Percentage of patients who survived more than 6 months from the date of surgery to death
Ratio of 12months overall survival (OS) | 12 months
  Percentage of patients who survived more than 12 months from the date of surgery to death
Progression-free survival (PFS) | 24 months
  Progression-free survival, time from the date of surgery to any types of progression
Overall survival (OS) | 24 months
  Overall survival, time from the date of surgery to death for whatever reason

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China